CLINICAL TRIAL: NCT06489678
Title: The Benefit of Cone-beam Computed Tomography and Robotic Assisted Bronchoscopy for the Diagnosis of Peripheral Pulmonary Lesions and Other Lung Disease Requiring Lung Biopsy: an Open-label, Randomized, Controlled Trial.
Brief Title: Benefit of Cone-beam CT and Robotic-assisted Bronchoscopy During Bronchoscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Thomas Gaisl, Sponsor Investigator, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BASEC Nr. 2024-00684
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Lung Neoplasms; Diagnosis; Lung Cancer
Keywords: Cone-beam CT; Robotic assisted Bronchoscopy; Cios Spin; Ion endoluminal System; Advanced Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Usual Care (No Intervention): For the control arm, standard bronchoscopy (±virtual or electromagnetic navigation, r-EBUS, and 2-dimensional fluoroscopy) will be employed, using various types of bronchoscopes (±ultra-thin bronchoscopes) and biopsy tools (needle, cryoprobe, forceps) at the investigator's discretion.
- Cone-beam CT and robotic assisted bronchoscopy (Active Comparator): Usual care with Cone-beam CT and the added option for the use of robotic assisted bronchoscopy (Ion endoluminal System, Intuitive) during the procedure. A connection between the cone-beam CT and the robotic system (NaviLink) is also possible.
  Interventions: Diagnostic Test: Robotic Assisted Bronchoscopy

INTERVENTIONS:
Diagnostic Test: Robotic Assisted Bronchoscopy — Cone-beam computed tomography (CBCT) technology and robotic-assisted bronchoscopy (RAB) present promising methods to enhance biopsy accuracy and procedural safety through 3-dimensional reconstructions and increased bronchoscope tip flexibility. Additionally, the transfer of navigational data between CBCT and RAB may further improve diagnostic yield. Given their distinct approaches to enhancing diagnostic outcomes, two separate study arms are warranted for CBCT and RAB.
  Other Names: Cios Spin (Siemens) and Ion endoluminal system (Intuitive)
  Arms: Cone-beam CT and robotic assisted bronchoscopy

SUMMARY:
This randomized controlled trial evaluates the integration of cone-beam computed tomography (CBCT) and robotic-assisted bronchoscopy (RAB) for diagnosing pulmonary lesions, hypothesizing improved diagnostic yield compared to traditional methods. The trial involves 2 study arms (2x46 lesions) over 24 months with 12 months of follow-up and the diagnostic yield (ATS 2024 criteria) as the primary endpoint.

DETAILED DESCRIPTION:
This randomized-controlled-trial, classified as Category A under Art 6 ClinO-MD, investigates the potential benefits of integrating cone-beam computed tomography (CBCT) and robotic-assisted bronchoscopy (RAB) into clinical practice for diagnosing pulmonary lesions. The study aims to enhance biopsy accuracy and safety by utilizing 3-dimensional reconstructions and increased flexibility of the bronchoscope tip. It targets two main clinical scenarios: peripheral lung lesions (PPLs) and other lung diseases requiring tissue biopsies. The hypothesis is that CBCT and RAB will significantly improve diagnostic yield compared to traditional 2D fluoroscopy techniques and endobronchial ultrasound.

The trial will involve 300 participants in the overall observational study, with a nested randomized controlled trial (RCT) for specific lesion types, targeting 2x46 lesions for 2 study arms i) usual care, ii) CBCT and RAB .

Primary endpoints include procedure time for the overall trial and diagnostic yield (ATS 2024 criteria) for the nested RCTs, analyzed via Pearson's Chi-squared test and multivariable logistic regression. Inclusion criteria encompass patients aged 18 or older, scheduled for bronchoscopy, with necessary pre-interventional exams and informed consent. Exclusion criteria include inability to tolerate the procedure, pregnancy, previous trial randomization, and specific lung conditions. The study's recruitment phase spans 24 months, with a 12-month follow-up, running from July 2024 to July 2027.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* Scheduled for bronchoscopy in order to obtain at least 1 specimen(s) of the lung via transbronchial biopsy
* Necessary periinterventional laboratory examinations and other examinations needed for the bronchoscopy
* Informed consent

Exclusion Criteria:

* Not able to tolerate procedure (bronchoscopy or apnea for CBCT)
* Previous randomization to an arm of the present trial
* Endobronchial lesion causing lobar atelectasis
* Inability or contraindications to undergo bronchoscopy (e.g. severe cardiopulmonary diseases, coagulation disorders, intolerance to anesthesia or endoscopic operation, psychiatric disorders, or severe neurosis)
* Pregnant or lactating women

For nested RCTs (Trial A + B):

* A: At least 1 peripheral lung lesion suspicious for lung cancer, beyond the visual range of the bronchoscope, rounded or irregular opacity, may be well or poorly defined, measuring ≤3 cm in diameter of the short axis (in CT scan)
* B:At least 1 peripheral target lung lesion of any kind beyond the visual range of the bronchoscope (measuring >3 cm in diameter of the short axis and/or with an interstitial pattern)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield | Including a 12-month follow-up (clinical data)
  ATS 2024 consensus criteria

SECONDARY OUTCOMES:
Radiation exposure | During Intervention
  Dose area product
Safety profile | During Intervention
  Rates of complications (bleeding, pneumothorax, pneumonia)
Diagnostic accuracy for milignancy | Including a 12-month follow-up (clinical data)
  True positives + true negatives / true positives + true negatives + false positives + false negatives
Quality of biopsies | During Intervention
  Number of malignant cells, suitability rates for further molecular pathological testing
Navigation success | During Intervention
  Anatomical confirmation of the position of the catheter in front or within the lesion as confirmed by r-EBUS or CBCT [not fluoroscopy]

OTHER OUTCOMES:
Procedure Duration | During Intervention
  Time of the whole procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gaisl, MD MPH PhD, Study Director — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No